CLINICAL TRIAL: NCT02841124
Title: Decision to Limit or Withdraw Specific Therapies for Advanced Cancer and Hematological Malignancies : Physicians and Patients Points of View and Interactions.
Brief Title: Decision to Limit or Withdraw Specific Therapies for Advanced Cancer and Hematological Malignancies.
Acronym: WHATELSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Saint Antoine, Paris (Unknown); Centre de Lutte Contre le Cancer Alexis Vautrin, Vandoeuvre les Nancy (Unknown); Centre Hospitalier de Colmar (Other); Clinique Devron, Dijon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: WHATELSE
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Cancer; Ethics
Keywords: Decision making
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Qualitative research (Other): Semi-structured interviews
  Interventions: Other: interviews

INTERVENTIONS:
Other: interviews — face-to-face interviews with the referent oncologist (or hematologist) and his patient (conducted by a physician and a psychologist respectively) as well as interviews with other partners involved in the situation (care staff and relatives)

SUMMARY:
The decision to limit or withdraw specific therapies (DLWT) in patients with advanced cancer is a complex process that is always painful for patients, relatives and professionals. For more than 10 years, shared decision making has been more and more emphasized. However, few data in the literature rely on clinical research. In order to understand their difficulties and issues, this study explores the determinants and modalities of DLWT and analyses the feasibility of different methods for investigating this decision making process.

DETAILED DESCRIPTION:
This study explores the decision-making process for patients with advanced cancer when the question to imit or withdraw specific therapies (DLWT) is raised, with a cross-analysis of physicians and pts points of view.

This study took place in 5 oncology and hematology units : 2 university hospitals, 1 general hospital, 1 cancer center and 1 private hospital. The study included two different approaches: an epidemiological section to identify the prevalence of these situations in different institutions and a qualitative study section exploring factors influencing the decision process. The epidemiological analysis included all hospitalized patients identified with advanced cancer for whom the question of DLWT was raised in a given week or during the two weeks preceding the investigation.

The qualitative analysis was based on interviews with the referent oncologist (or hematologist) and his patient (conducted by a physician and a psychologist respectively) as well as interviews with other partners involved in the situation (care staff and relatives) depending on the center. Researchers also participated in multidisciplinary meetings and monitored changes in the decision over a three month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cancer
* Existence of a questioning about DLWT
* Absence of guide lines

Exclusion Criteria:

* Incapacity of the patient to participate to an interview
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
interviews with physicians, patients and relatives | 6 months
  A thematic analysis induces the creation of a set of themes and concepts clustered by relevance into a tree structure. The thematic tree structure constitutes the dataset of interest.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier de Colmar, Colmar
  - Clinique Drevon, Dijon
  - Centre Hospitalier Universitaire St Antoine, Paris
  - Centre de Luttre Contre le Cancer Alexis Vautrin, Vandœuvre-lès-Nancy